CLINICAL TRIAL: NCT02035943
Title: Tight Glycemic Control and Insulin Administration During Parenteral Nutrition, in Critical Ill Patients
Brief Title: Tight Glycemic Control and Insulin Administration During Parenteral Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 127
Record Dates: First submitted 2011-12-01; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Critical Ill Patient Undergone Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin separated (Active Comparator): Seprated infusion of insulin
  Interventions: Dietary Supplement: Insulin separated
- Insulin added to parenteral nutrition (Active Comparator): Insulin added to parenteral nutrition
  Interventions: Dietary Supplement: Insulin added to parenteral nutrition

INTERVENTIONS:
Dietary Supplement: Insulin separated — separate continuos infusion of insulin
  Arms: Insulin separated
Dietary Supplement: Insulin added to parenteral nutrition — Insulin added to parenteral nutrition
  Arms: Insulin added to parenteral nutrition

SUMMARY:
In this study the investigators want to comare safety and efficacy of two different metods to administrate insulin during parenteral nutrition.

DETAILED DESCRIPTION:
In this study the investigators want to compare safety and efficacy of two different metods to administrate insulin during parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Critical ill patients undergone parenteral nutrition

Exclusion Criteria:

* Acute cerebral injury, pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number of glucose level control out of range (80-110 mg/dl) | ICU stay (a week on average)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio De Chiara, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, MI, Italy